CLINICAL TRIAL: NCT00457171
Title: A Double-Blind, Placebo-Controlled Phase I/II Study in Patients With Mild to Moderate Ulcerative Colitis Treated With GI-270384X, an Oral ICAM-1 and E-Selectin Inhibitor
Brief Title: GI-270384 Study In Patients With Mild To Moderate Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: EBD100729
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Ulcerative Colitis
Keywords: GI-270384 colitis patients ECAM oral
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Drug: GI-270384

SUMMARY:
The aim of this double blind, placebo controlled, study is to evaluate activity consistent with efficacy provided by 14 days administration of GI270384X, and to provide preliminary pharmacokinetics and safety/tolerability of 14 days administration of GI270384X in patients with mild to moderate active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion criteria:

* Females can be of childbearing or non-childbearing potential
* Subjects who have relapsing (relapsed = 6 weeks ago; this being at least a second episode) mild to moderate UC (score of 4 - 11 on the MTWI at Screening and with an endoscopy score of = 2). Diagnosis of UC originally must be established by sigmoidoscopy or colonoscopy, and have compatible histology.
* As confirmed through signed informed consent, the subject must understand and be able, willing and likely to fully comply with study procedures and restrictions

Exclusion criteria:

* Subjects with severe UC according to the MTWI (score >11) and subjects who have been in relapse for > 6 weeks.
* Subjects are not eligible for this study if they have Crohn's Disease, proctitis (where the extent of inflammation = 15 cm), bleeding disorders, or active ulcer disease.
* Positive stool culture for enteric pathogens (including Salmonella, Shigella, Yersinia, Aeromonas, Plesiomonas or Campylobacter).
* Presence of Clostridium difficile toxin present or with ova or parasites as detected by microscopy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2004-12

PRIMARY OUTCOMES:
Modified Truelove/Witts activity index for disease severity, between baseline and week 4 Endoscopic severity at 2 weeks Quality of life, as assessed by Inflammatory Bowel Disease Questionnaire, and changes on UC imaging scanning (leukocyte scan)

SECONDARY OUTCOMES:
Vital signs (blood pressure, heart rate, body weight, 12-lead ECG), clinical laboratory data (haematology, clinical chemistry, urinalysis) and adverse events Cmax and AUC(0-4) of GI270384X, GI266193X and GW277348X after 14 days dosing.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, B.Sc., Study Director — GlaxoSmithKline